CLINICAL TRIAL: NCT04178226
Title: The Comparison of Efficacy of Manual Acupuncture and Laser Acupuncture on Autonomic Nervous Activity and Quality of Life in Women With Dysmenorrhea.
Brief Title: The Efficacy of Two Types of Acupuncture on Autonomic Nervous Activity and Quality of Life in Women With Dysmenorrhea.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TCHIRB-10712112
Record Dates: First submitted 2019-11-19; First posted 2019-11-26 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Dysmenorrhea
Keywords: acupuncture; laser acupuncture; Autonomic nerve activity; dysmenorrhea; prostaglandin; quality of life
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: 1. Control group
  2. Acupuncture group
  3. Laser acupuncture group Patients in acupuncture/ laser acupuncture group will be crossover to another group after 3 courses of treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): conventional therapy (NSAIDs and OCP)
- Manual Acupuncture (Experimental): manual acupuncture therpy
  Interventions: Other: Manual Acupuncture
- Laser Acupuncture (Experimental): laser acupuncture therapy
  Interventions: Device: Laser Acupuncture

INTERVENTIONS:
Other: Manual Acupuncture — The acupoints choose are (RN6) (RN4) (SP6) (PC6) (SP10) (SP4)
  Arms: Manual Acupuncture
Device: Laser Acupuncture — The acupoints choose are (RN6) (RN4) (SP6) (PC6) (SP10) (SP4)
  Arms: Laser Acupuncture

SUMMARY:
Integrative medicine raises public's attention due to either mainstream or traditional medicine has its limitation. The topic "dysmenorrhea", with prevalence up to 50%, troubled many females with symptom as depression, reduced the quality of life; and even withdraw from daily activity.

Clinically, gynecologists apply analgesic such as Non-steroidal Anti-inflammatory Drugs, and oral contraceptive pills or progestin as conventional therapy. As NSAIDs cause gastrointestinal discomfort, while hormone therapy leads to other concerns; some women now adopt acupuncture as an alternative therapy for its safety.

Furthermore, laser acupuncture has been practiced in recent years for it integrates the meridian theory and laser therapy; hence there are also some positive research in academic field.Whether laser or traditional acupuncture is more effective is still under debate.

Additionally, investigators had published that the theory of yin/yang (meridian) is compatible with autonomic nerve theory. As many women with dysmenorrhea suffered from insomnia, anxiety, convulsion of the uterine muscle, which are related to autonomic nerve dysfunction, investigators are intrigued to know whether the effect of acupuncture is related to adjusting autonomic nerve system.

Investigators intend to investigate the efficacy of laser and manual acupuncture in dysmenorrhea, and whether their mechanism is germane to hormone alternation or autonomic nervous system adjustment. The points in this proposal are 1.evaluate the efficacy of manual/laser acupuncture in dysmenorrhea in respects of symptoms and quality of life 2. compare whether these types acupuncture will alter the prostaglandin or hormone and the relationship between with the efficacy. 3. evaluate whether the mechanism of manual and laser acupuncture is relevant to alternating the autonomic nerve activity and if not correspond to Yin-Yang theory.

DETAILED DESCRIPTION:
1.1 The prevalence and mechanism of dysmenorrhea Dysmenorrhea is a troubling problem affect more than 50% reproductive-aged women and affect females' quality of life is not only physical but also psychologic aspects. It costs a lot of health, social and economic burden. The symptom is characterized by cramping pain in the lower abdomen, starting within the first eight to 72 hours of menstruation. According to research, the severity of dysmenorrhea ranged widely from mild, tolerable to incapability for 1 to 3 days each menstrual cycle, even incapable of work or daily activity. Some women even suffer from autonomic dysfunction symptoms such as dizziness, diarrhea, migraine, vomiting, unable to concentrate, negative mood and anxiety or depression. The mechanism of pain associated with dysmenorrhea can be addressed by two aspects: neuro-endocrine regulated and neuro-physiologic related. One is by the action of prostaglandins such as prostaglandin E2, prostaglandin F2α, or vasopressin-related from the endometrium at the onset of menstruation which stimulates pain neurons and induces excessive contraction of the uterus. Prostaglandin production is controlled by progesterone: when progesterone levels drop, immediately prior to menstruation, prostaglandin levels increase. The other aspect is that the increasing uterine muscle contractions and hormone secretion is regulated by the sympathetic nervous system. Therefore, some scholars stress the importance of reducing sympathetic tone or re-imbalance the autonomic nervous activity. Accordingly, investigators note that some research such as yoga, or aerobic exercise applied in dysmenorrhea are designed through this approach.

1.2 Current treatment of dysmenorrhea The conventional treatments adopt the use of non-steroidal anti-inflammatory drugs (NSAIDs) combined with oral contraceptives or progestins. Hormonal contraceptives are the first-line treatment for dysmenorrhea caused by endometriosis. Topical heat, exercise, and nutritional supplementation may be beneficial in patients who have dysmenorrhea. The NSAIDs may induce gastrointestinal disturbance while the hormone treatment may increase the risk of some cancer or other heart problems; therefore, around 25% of patients are refractory to conventional therapy. Some women choose alternative therapies such as yoga, acupuncture, or massage for relieving their pain albeit the evidence of these therapies is not enough.

1.3 The role of acupuncture in dysmenorrhea Acupuncture, which is non-invasive and with few side effects; has been proved with well anesthetic effect in pain control through varied mechanisms. On one hand, some study propose that the mechanism of acupuncture in dysmenorrhea is based on changes in neurophysiologic and neuro-hormonal activities such as endogenous opioid, serotonin, and acetylcholine which results in pain reduction; on the other hand, some study indicate that acupuncture has an effect in the reduction of inflammation, alterations in uterine blood flow and changes in prostaglandin levels. Previous research confirmed that acupuncture affects the autonomic status to some extent in diverting circumstances, yet the style of acupuncture varied from manual to warm to laser acupuncture etc. In addition to pain relieving, acupuncture has been reported with the efficacy in improving the quality of life and decreasing NSAID use after regular treatment for 3 to 6 months.

1.4 manual acupuncture VS Laser acupuncture Laser acupuncture raises the public's attention for its much less invasive than real acupuncture. In previous time, only TCM doctors or acupuncturists could practice the acupuncture; yet since laser acupuncture is not invasive, mainstream (western medicine) physicians could also practice laser therapy in the clinic, more and more research about laser acupuncture was published in the field of pain control, orthopedics, and internal medicine. Nevertheless, the research regarding laser acupuncture applied in dysmenorrhea is rare, only one trial is noted in the Pubmed, which intrigues us to further investigate the potential effect of laser acupuncture in dysmenorrhea now that investigators already have abundant manual acupuncture experience in this issue. Additionally, it is believed that acupuncture could attenuate pain or improve microcirculation by regulating the autonomic nervous system. However, whether the effect of manual and laser acupuncture on autonomic nerve activity is the same is still controversial. Some study indicates laser acupuncture could be an alternative stimulate therapy for it has the same effect as manual acupuncture on vagal activity whereas still, other studies note laser acupuncture has a different effect from manual acupuncture on autonomic activity. As a result, investigators aim to know more about these two types acupuncture's effect on HRV and compare their effectiveness.

1.5 Prospective of laser acupuncture in dysmenorrhea As many females troubled with the dysmenorrhea and hormone or analgesics therapy has a certain effect, acupuncture is promising for its less-invasiveness. Furthermore, if laser acupuncture is non-inferior to manual acupuncture or even much more effective; then it could be another alternative therapy in this issue.

1.6 The correlation of Meridian system and Autonomic system in acupuncture study In recent decades, more and more researchers demonstrated that the meridian system corresponds to the nervous system or has some overlapping with it. The study indicated that stimulating some acupoints or meridians could change the autonomic activity and attain the goal of improving some physiologic problem. Chien et al in 2014 indicated that acupoints stimulation could modulate the autonomic nervous system to exert its physiological effect through the pathway of the meridian system. Cui et al revealed that stimulating Heart Meridian may improve AMI by inhibiting sympathetic discharges and elevating vagal discharges in AMI rats. These studies confirmed the relationship between meridian and autonomic system, yet few studies compare the efficacy or mechanism of different treatments (medication or different types acupuncture) in applying in the same disease. That is why investigators intend to apply two different acupuncture (manual and laser) to compare their effect on autonomic nervous system and efficacy in clinics.

1.7 Autonomic nerve activity V.S manual/ laser acupuncture V.S dysmenorrhea As has mentioned, acupuncture works through regulating yin-yang and meridian energy. The interesting thing is that from our previous study, investigators found that the concept of parasympathetic/sympathetic system is compatible with yin/yang theory in Chinese Medicine to a certain extent; while the promotion of energy is consistent with the "De-Qi" in performing acupuncture. Since the symptoms related to dysmenorrhea such as pain, diarrhea, headache, poor sleep are also related to autonomic dysfunction. (imbalance of sympathetic/parasympathetic tone); investigators are intrigued by whether the mechanism of acupuncture is relevant to the improvement of autonomic nerve activity in dysmenorrhea. Do the manual and laser acupuncture work through the same mechanism on autonomic nerve system or meridian network? Accordingly, under the context that acupuncture might have an effect on reconciling the autonomic nervous imbalance and yin/yang in dysmenorrhea and to further understand this issue, investigators intend to compare the manual, laser acupuncture and conventional treatment reflecting in autonomic nervous activity and effect on dysmenorrhea.

1.8 The relationship of hormone and dysmenorrhea Previous research noted that the dysmenorrhea may be caused by the overproduction of uterine prostaglandins (PGs), which might be regulated by progesterone, though not totally depend only on endocrine factors. All women have increased levels of PGs during the luteal phase compared with the follicular phase of ovulatory cycles. However, compared with eumenorrheic women, dysmenorrhea women have higher levels of PGs and the concentration of progesterone per menstruation was significantly higher in the eumenorrheic women than in the dysmenorrhea patients as well. Some gynecologists even use prostaglandin synthetase inhibitor ( ex. Ibuprofen) in dealing with the dysmenorrhea. The shift of estradiol/progesterone ratio in favor of estradiol contributes to the underlying pathogenic principle of dysmenorrhea. Therefore, the change of hormones could present the level of improvement of dysmenorrhea.

2.1 Acupuncture applied in dysmenorrhea From research, acupuncture is very popular when it comes to some gynecologic problems, such as menopause symptoms or premenstrual syndrome. However, most study focus on the comparison of acupuncture and sham acupuncture or NSAID and the acupuncture protocol is not conclusive; some chose only one acupoint (SP6) while others chose a group of acupoints. So far, none of the studies compares the efficacy and effect on HRV or changes on hormone and prostaglandin between in manual and laser acupuncture.

2.2 Heart rate variation (HRV) VS Cytokine and Acupuncture Regarding the connection of acupuncture and autonomic nerve system or Heart rate variation (HRV), Acupuncture is hypothesized to modulate the neuroendocrine and autonomic nervous system and thereby revitalize the balance of metabolism in the body. Investigators noted some evidence confirmed that acupuncture could improve depression, fatigue through regulating cytokine and autonomic nervous system. Nevertheless, whether there will be any relationship between the cytokine change and HRV activity is uncertain. As a result, the study is designed for checking the correlation of change in cytokine (Prostaglandin, estrogen, progesterone) and HRV activity in dysmenorrhea beyond the evaluation of comparing efficacy. Investigators suppose the phenomenon of decreased prostaglandins and increased progesterone will be noted in dysmenorrhea patients benefit from acupuncture.

The investigators design not only aim to compare the efficacy of manual, laser acupuncture and control group in dysmenorrhea but also further investigate whether their effect on HRV is different. The acupoints investigators chose are most located in Yin meridians which correspond to Yin-Yang theory that " Yang masters Chi while Ying masters blood "and "Yang is frequently in excess while yin is often in deficiency". Investigators aim to reconcile the yin-yang through the special designed acupoints protocol. Additionally, investigators can also confirm whether the effect of manual and laser acupuncture in dysmenorrhea is related to the improvement of autonomic nerve activity and try to integrate our understanding about neurophysiology and acupuncture along with TCM-Yin/Yang theory based on the previous study. Whether acupuncture could change the hormone peptides or cytokine would be evaluated to clarify the mechanism of how manual or laser acupuncture work. Investigators expect the study can promote the crosstalk between the Chinese and western medicine and provide more definitive evidence for acupuncture applied in dysmenorrhea.

Objective and approach Investigators design a three-arms clinical randomized study, which includes manual acupuncture, laser acupuncture and conventional therapy (NSAIDs and OCP) and enrolls women with dysmenorrhea.

Specific Aims Specific aim 1: To compare the efficacy of manual and laser acupuncture and control group (conventional therapy: including NSAIDs) in dysmenorrhea.

Specific aim 2:To evaluate whether the laser and manual acupuncture will affect the serum prostaglandin, and hormone and the relationship between with the efficacy in dysmenorrhea.

Specific aim3: To identify the relationship between autonomic nerve activity change and laser / manual acupuncture reflect in dysmenorrhea and integrate with the TCM -Yin/Yang and meridian theory.

ELIGIBILITY:
Inclusion Criteria:

1. Women within reproductive age (15 to 49 years);
2. Participants who complain about dysmenorrhea with at least grade II level.
3. Self-reported lower abdominal and pelvic, medial anterior thigh pain or low back pain associated with the onset of menses and lasting in 72 hours.
4. Some accompanied symptoms as dizziness and syncope, cramping, nausea, vomiting, diarrhea, headaches, and fatigue present compatible with the menses cycle were also included.

Exclusion Criteria:

1. Dysmenorrhea resulting from the use of an intra-uterine device (IUD);
2. Mild or infrequent dysmenorrhea.
3. Dysmenorrhea with possible underlying tumor or malignancy

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
The serum prostaglandin E2 level change. | baseline, after 3 months treatments, after 1 month wash out, after another 3 months treatments
  serum test
The autonomic nerve activity change. | baseline, before and after every month treatment for 3 months, after 1 month wash out, before and after every month treatment for 3 months.ts
  Heart rate variance equipment

SECONDARY OUTCOMES:
The quality of life change. | baseline, after every month treatment for 3 months, after 1 month wash out, after every month treatment for 3 months.ts
  SF-12 quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tsai-Ju Chien, PhD, Study Chair — Taipei City Hospital
Locations (1):
- Taipei City Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Iacovides S, Avidon I, Bentley A, Baker FC. Reduced quality of life when experiencing menstrual pain in women with primary dysmenorrhea. Acta Obstet Gynecol Scand. 2014 Feb;93(2):213-7. doi: 10.1111/aogs.12287. Epub 2013 Nov 25. PMID 24266425
- [Background] Bernardi M, Lazzeri L, Perelli F, Reis FM, Petraglia F. Dysmenorrhea and related disorders. F1000Res. 2017 Sep 5;6:1645. doi: 10.12688/f1000research.11682.1. eCollection 2017. PMID 28944048
- [Background] Hasegawa N. [Dysmenorrhea and the autonomic nervous system]. Sanfujinka No Jissai. 1968 Jun;17(6):492-8. No abstract available. Japanese. PMID 5755245
- [Background] Osayande AS, Mehulic S. Diagnosis and initial management of dysmenorrhea. Am Fam Physician. 2014 Mar 1;89(5):341-6. PMID 24695505
- [Result] Smith CA, Zhu X, He L, Song J. Acupuncture for primary dysmenorrhoea. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD007854. doi: 10.1002/14651858.CD007854.pub2. PMID 21249697
- [Result] Taguchi R. Acupuncture anesthesia and analgesia for clinical acute pain in Japan. Evid Based Complement Alternat Med. 2008 Jun;5(2):153-8. doi: 10.1093/ecam/nem056. PMID 18604250
- [Result] McDonald JL, Cripps AW, Smith PK. Mediators, Receptors, and Signalling Pathways in the Anti-Inflammatory and Antihyperalgesic Effects of Acupuncture. Evid Based Complement Alternat Med. 2015;2015:975632. doi: 10.1155/2015/975632. Epub 2015 Aug 3. PMID 26339274
- [Result] Stener-Victorin E, Waldenstrom U, Andersson SA, Wikland M. Reduction of blood flow impedance in the uterine arteries of infertile women with electro-acupuncture. Hum Reprod. 1996 Jun;11(6):1314-7. doi: 10.1093/oxfordjournals.humrep.a019378. PMID 8671446
- [Result] Witt CM, Reinhold T, Brinkhaus B, Roll S, Jena S, Willich SN. Acupuncture in patients with dysmenorrhea: a randomized study on clinical effectiveness and cost-effectiveness in usual care. Am J Obstet Gynecol. 2008 Feb;198(2):166.e1-8. doi: 10.1016/j.ajog.2007.07.041. PMID 18226614
- [Result] Kempf D, Berger D, Ausfeld-Hafter B. [Laser needle acupuncture in women with dysmenorrhoea: a randomised controlled double blind pilot trial]. Forsch Komplementmed. 2009 Feb;16(1):6-12. doi: 10.1159/000193294. Epub 2009 Feb 4. German. PMID 19295224
- [Result] Shu Q, Wang H, Litscher D, Wu S, Chen L, Gaischek I, Wang L, He W, Zhou H, Litscher G, Liang F. Acupuncture and Moxibustion have Different Effects on Fatigue by Regulating the Autonomic Nervous System: A Pilot Controlled Clinical Trial. Sci Rep. 2016 Nov 25;6:37846. doi: 10.1038/srep37846. PMID 27886247
- [Result] Wu JH, Chen HY, Chang YJ, Wu HC, Chang WD, Chu YJ, Jiang JA. Study of autonomic nervous activity of night shift workers treated with laser acupuncture. Photomed Laser Surg. 2009 Apr;27(2):273-9. doi: 10.1089/pho.2007.2235. PMID 18785846
- [Result] Wong YM. Effect of Laser Acupuncture on Heart Rate Variability of Nonpatients and Patients with Spinal Cord Injury. J Acupunct Meridian Stud. 2017 Jan;10(1):53-54. doi: 10.1016/j.jams.2016.11.004. Epub 2016 Nov 29. PMID 28254104
- [Result] Chien LW, Chen FC, Hu HY, Liu CF. Correlation of electrical conductance in meridian and autonomic nervous activity after auricular acupressure in middle-aged women. J Altern Complement Med. 2014 Aug;20(8):635-41. doi: 10.1089/acm.2012.0900. Epub 2014 May 27. PMID 24865945
- [Result] Litscher G. Bioengineering assessment of acupuncture, Part 6: monitoring--neurophysiology. Crit Rev Biomed Eng. 2007;35(1-2):1-36. doi: 10.1615/critrevbiomedeng.v35.i1-2.10. PMID 17956221
- [Result] Schmidt K. [Should acupuncture be reimbursable? Yin and yang in significant conflict]. MMW Fortschr Med. 2000 Aug 24;142(33-34):52. No abstract available. German. PMID 10998908
- [Result] Larroy C. Comparing visual-analog and numeric scales for assessing menstrual pain. Behav Med. 2002 Winter;27(4):179-81. doi: 10.1080/08964280209596043. PMID 12165972
- [Result] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Derived] Chien TJ, Chang YI, Liao LL, Hsu YN, Huang CW. Comparative Efficacy of Low-Level Laser Acupuncture and Electroacupuncture in Women With Dysmenorrhea and Autonomic Imbalance: A Pilot Randomized-Controlled Trial. Pain Res Manag. 2025 Oct 23;2025:3494216. doi: 10.1155/prm/3494216. eCollection 2025. PMID 41179650
- [Derived] Chien TJ, Huang YS, Liao LL, Chu CC, Pai JH. Head-to-Head Comparison of Electroacupuncture and Laser Acupuncture Effects on Autonomic Regulation and Clinical Effects in Dysmenorrhea: A Randomized Crossover Clinical Trial. J Integr Complement Med. 2024 Jun;30(6):560-575. doi: 10.1089/jicm.2023.0183. Epub 2024 Feb 16. PMID 38364185